CLINICAL TRIAL: NCT04481399
Title: mHealth Tools to Improve Service Delivery Quality of an Evidence-Based Family Home Visiting Intervention to Prevent Family Violence Among High Risk Families in Sierra Leone
Brief Title: Mobile Health (mHealth) Tools to Improve Delivery Quality of a Family Home Visiting Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: Caritas Freetown (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alethea Desrosiers, Research Assistant Professor, Boston College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21.006.01; R21MH124071 (NIH)
Record Dates: First submitted 2020-07-15; First posted 2020-07-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Parent-Child Relations; Behavioral Intervention; Exposure to Violent Event; Child Development; Mental Health; Implementation Science; mHealth; Community Health Workers
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FSI-ECD (Experimental): The Family Strengthening Intervention for Early Childhood Development (FSI-ECD) is an evidence-based home-visiting behavioral intervention for vulnerable families with children aged 6-36 months. The FSI-ECD targets improving parental emotion regulation and parent-child interactions to improve parental mental health and child development outcomes and reduce family violence. The FSI-ECD will be delivered in weekly 90-minute home visiting sessions for 12 consecutive weeks.
  Interventions: Behavioral: Family Strengthening Intervention for Early Childhood Development
- Control (Other): The control is standard maternal and child health home visiting delivered by community health workers. Families will receive three 90-minute home visiting educational sessions focused on nutrition, hygiene, and post-natal care.
  Interventions: Other: Community Health Worker Routine

INTERVENTIONS:
Behavioral: Family Strengthening Intervention for Early Childhood Development — The Family Strengthening Intervention for Early Childhood Development (FSI-ECD) is an evidence-based home-visiting behavioral intervention for vulnerable families with children aged 6-36 months. The FSI-ECD targets improving parental emotion regulation and parent-child interactions to improve parental mental health and child development outcomes and reduce family violence. FSI-ECD compromises five core components delivered in 12 modules delivered in weekly sessions via active coaching by community health workers. Core components include coaching on: a) nutrition, health and hygiene; b) early stimulation and playful parenting; c) building resilience and coping skills; d) building problem-solving skills; and d) building emotion regulation and conflict resolution skills.
  Arms: FSI-ECD
Other: Community Health Worker Routine — Standard CHW care involves three home visiting sessions delivered to families following childbirth with weekly supervision via phone or face-to-face. Topics of home visiting sessions include: skilled post-natal care for mothers, early initiation of breastfeeding and exclusive breastfeeding practices, adequate nutrition, immunization services and timely use of these services, hand washing and hygiene practices (including waste disposal and food hygiene), building the capacity of family members to appropriately take care of newborns and children under age 5, and building the capacity of family members to recognize and act on postnatal danger signs for newborns, mothers, and children under 5. CHWs also conduct screenings for acute malnutrition and growth monitoring to identify early referrals, and they can provide family planning methods, deworming tablets and other vitamins for acute malnutrition, dehydration, and anti-malaria treatment. Each home-visiting session lasts about 60 minutes.
  Arms: Control

SUMMARY:
This study will pilot a family-focused, behavioral health intervention while also developing and piloting mHealth tools to support Community Health Workers (CHWs) in Sierra Leone. This dual focus will help build capacity both for delivery of evidence-based mental health services to reduce family violence and harsh parenting practices, and for effective use of mHealth strategies to improve healthcare delivery quality. This study will leverage Government of Sierra Leone investments in community health initiatives as a strategy to address critical healthcare workforce limitations that plague delivery of evidence-based interventions to vulnerable families in post-conflict Sierra Leone. Study aims are to:

Aim 1. Employ a five-phase user-centered design approach to develop and test mHealth tools to improve training, supervision, and fidelity monitoring of Community Health Workers. Study investigators hypothesize that mHealth tools will be feasible, acceptable, and user-friendly.

Aim 2. Conduct a Randomized Controlled Pilot Study to assess feasibility, acceptability, costs and preliminary effects of the mHealth-supported delivery of FSI-ECD on parent mental health, emotion regulation, and familial violence in high risk families with children aged 6-36 months (n=40) in comparison to control families (n=40) who receive standard care. Parental mental health, emotion regulation, household violence, and parenting practices will be assessed at baseline, post-intervention and 6-month follow-up. Study investigators hypothesize that (a) the effects of the FSI-ECD will be comparable to results observed with vulnerable families in Rwanda; (b) digital tools will be feasible and acceptable to CHWs and supervisors.

Aim 3. Leverage well-established relationships and government partners to strengthen capacity for mHealth research and quality healthcare delivery in Sierra Leone. Partners include the University of Makeni, the Directorate of Science, Technology and Innovation, and the Ministry of Health and Sanitation.

ELIGIBILITY:
Inclusion Criteria:

* Focus Group-User Interface/User Experience (UI/UX) Participants: Aged 18 or older; ability to attend 1-2 sessions (90 minutes per session)
* Family Participants: Families who are (a) a Sierra Leonean household with cohabitating caregivers (e.g., father/mother, mother/grandmother, mother/intimate partner), and child (aged 6-36 months) with both parents aged 18 or older and; (b) one parent scoring at least 62.5 on the Difficulties in Emotion Regulation Scale (DERS). The DERS cut-off score has been used successfully as a risk assessment screening tool in our prior and ongoing studies in Sierra Leone. Sierra Leonean caregivers scoring above this threshold on the DERS have reported significantly higher levels of severe physical punishment with their children as well as intimate partner violence. Both parents must agree to attend FSI-ECD sessions. If enrolled families have more than one child aged 6-36 months, we will include all eligible children as study participants.
* Community Health Worker Participants: CHWs who are 18 years or older and who are assigned to the Peripheral Health Unit that provides health services in one of our target communities.
* Community Health Worker Supervisor Participants: Supervisors are 18 years or older and oversee CHWs providing maternal and child health services

Exclusion Criteria:

* Focus Group-User Interface/User Experience (UI/UX) Participants: Individuals younger than age 18 and individuals who do not meet inclusion criteria.
* Family Participants: Families who do not meet all inclusion criteria and/or who are experiencing active family crises (e.g., current suicidality or psychosis, cognitive impairment, ongoing divorce process).
* Community Health Worker Participants: Individuals under age 18 cannot be recruited to work as a CHW.
* Community Health Worker Supervisor Participants: Individuals under age 18.

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed through the John Hopkins Implementation and Dissemination Science Scale | Immediately after the intervention
  Feasibility of mHealth tool implementation to support FSI-ECD delivery will be assessed via a Dissemination and Implementation measures developed by the John Hopkins Bloomberg School of Health. This is a 20-item self-report measure and items are scored on a 4-point Likert scale: 1=not at all, 2=a little bit, 3=a moderate amount, 4=a lot.
Acceptability as assessed through the John Hopkins Implementation and Dissemination Science Scale | Immediately after the intervention
  Acceptability of mHealth tool implementation to support FSI-ECD delivery will be assessed via a Dissemination and Implementation measures developed by the John Hopkins Bloomberg School of Health. This is a 10-item self-report measure and items are scored on a 4-point Likert scale: 1=not at all, 2=a little bit, 3=a moderate amount, 4=a lot.

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) | Baseline, immediately after the intervention, and 3-months after the intervention
  The Difficulties in Emotion Regulation Scale (DERS) is a 36-item measure that assesses emotion dysregulation across 6 domains, i.e., non-acceptance of emotional responses, difficulty engaging in goal-directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity. The DERS is scored on a 5-point Likert scale: 1=Almost Never, 2=Sometimes, 3=About half the time, 4=Most of the time, 5=Almost always. Higher scores indicate greater difficulties in emotion regulation.
Conflict Tactics Scale-2 (CTS-2) | Baseline, immediately after the intervention, and 3-months after the intervention
  The Conflict Tactics Scale (CTS-2) is a 78-item scale (39 behaviors or experiences, each asked once for respondent and one for partner). The CTS is comprised of 5 subscales, i.e., negotiation, psychological aggression, physical assault, injury, and sexual coercion. The response categories gauge the frequency with which acts were used during conflict with a partner in the past year using a 6-point scale ranging from "never" to "20 or more times." There are also response options of "Never in the last year, but it did happen before that," and "This has never happened."
Home Observation for Measurement of the Environment (HOME) | Baseline, immediately after the intervention, and 3-months after the intervention
  The Home Observation for Measurement of the Environment (HOME) is a 43-item measure that assesses the level of stimulation and support provided by caregivers in the home. All items receive a binary score based on the presence (score = 1) or absence (score = 0) of self-reported and direct observation of parenting behaviors and household conditions. Item scores are summed to derive scores on a total scale and the 6 subscales, i.e., variety, organization, acceptance, involvement, learning materials, and responsivity.
Observation of Mother-Child Interaction (OMCI) | Baseline, immediately after the intervention, and 3-months after the intervention
  The Observation of Mother-Child Interaction (OMCI) is a direct observational measure used to assess mother-child interaction during a shared picture-book reading activity that includes maternal (10 items) and child assessments (5 items). Maternal responsive behaviors include contingent responding, emotional-affective support, support for infant foci of attention, and language inputs. Child behaviors include the child's behavioral and social-emotional reactions during the observation. Each item is rated on a 4-point scale: 0 = Never, 1 = Very few, 2 = Sometimes (3-4 times), and 3 = Five or more times. Total scores are assigned for the mother's reaction, the child's reaction, and mother-child interaction, respectively.
Hopkins Symptom Checklist (HSCL) | Baseline, immediately after the intervention and 3-months after the intervention
  The Hopkins Symptom Checklist (HSCL) is a 25-item inventory that measures symptoms of anxiety and depression. Part I of the measure has 10 items assessing anxiety symptoms and Part II has 15 items assessing depression symptoms. Each item is rated on a 4-point scale: 1 = Not at all, 2 = A little, 3 = Quite a bit, and 4 = Extremely. Item scores are summed to derive scores for the total scale and subscales, i.e., anxiety and depression.
Post-traumatic Stress Disorder Civilian Checklist | Baseline, immediately after the intervention and 3-months after the intervention
  The Post-traumatic Stress Disorder Civilian Checklist is a 17-item scale that assesses symptoms of Post-traumatic Stress Disorder. Items are rated on a binary scale of "yes" or "no" responses.

CONTACTS AND LOCATIONS:
Overall Officials: Alethea Desrosiers, PhD, Principal Investigator — Boston College
Locations (1):
- University of Makeni, Makeni, Sierra Leone

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be in accordance with the NIH Data Sharing Policy and Implementation Guidance and more specifically the "Data Sharing Expectations for National Institute of Mental Health (NIMH)-funded Clinical Trials". The data generated in this study will be entered into the NIMH Data Archive as required and prescribed by the Notice of Award as well as presented at national and/or international conferences and published in a timely fashion. All final peer-reviewed manuscripts that arise from this proposal will be submitted to the digital archive PubMed Central. Published data will be available in print or electronically from publishers, subject to subscription or printing charges. Research data that document, support and validate research findings will be made available after the main findings from the final research data set have been accepted for publication.
Time Frame: Data will become available after the main findings from the final research data set have been accepted for publication and will be available for 3 years following closeout of the award.
Access Criteria: The data generated in this clinical will be entered into the NIMH Data Archive as required and prescribed by the Notice of Award as well as presented at national and/or international conferences and published in a timely fashion. All final peer-reviewed manuscripts that arise from this proposal will be submitted to the digital archive PubMed Central. Published data will be available in print or electronically from publishers, subject to subscription or printing charges. Research data that document, support and validate research findings will be made available after the main findings from the final research data set have been accepted for publication.

REFERENCES:
- [Derived] Desrosiers A, Schafer C, Esliker R, Jambai M, Betancourt T. mHealth-Supported Delivery of an Evidence-Based Family Home-Visiting Intervention in Sierra Leone: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2021 Feb 2;10(2):e25443. doi: 10.2196/25443. PMID 33528371